CLINICAL TRIAL: NCT07269665
Title: A First-In-Human, Open Label, Dose Escalation Trial to Evaluate the Safety, Tolerability and Pharmacodynamics of a Single Dose of AXV-101 in Patients With Bardet-Biedl Syndrome 1 (BBS1) Bi-Allelic Mutations and Retinal Degeneration
Brief Title: First-in-Human, Dose Escalation Trial of AXV-101 in BBS1-Related Retinal Degeneration
Acronym: AXIS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Axovia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLIN101-AXV-101(SR); ISRCTN96250868 (Other: The UK's Clinical Study Registry)
Record Dates: First submitted 2025-09-16; First posted 2025-12-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bardet-Biedl Syndrome 1; Retinal Degeneration
Keywords: bi-allelic mutations; retinal degeneration; first-in-human; Bardet-Biedl syndrome 1; BBS1; gene therapy; children
MeSH Terms: conditions — Bardet-Biedl syndrome 1; Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: The study consists of two parts (cohort 1 and cohort 2). Cohort 1 will include up to three participants. Participants in this cohort will be administered a minimally effective dose of AXV-101 (3 E11 Viral genomes; Vg). The safety data for the first participant will be reviewed by an Independent Data Monitoring Committee (IDMC) before the next participants are enrolled. The IDMC will then review the next two participants' data before opening the next part of the study (Cohort 2).
  Cohort 2 will include up to nine participants. Participants in this cohort will be administered a therapeutic dose of AXV-101 (5 E11 Vg). The IDMC will review the safety data after each dose for the first three participants, and if no safety concerns are raised, the remaining six participants in cohort 2 will be dosed sequentially.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will include up to three participants. Participants in this cohort will be administered a minimally effective dose of AXV-101 (3 E11 Viral genomes; Vg). The safety data for the first participant will be reviewed by an Independent Data Monitoring Committee (IDMC) before the next participants are enrolled. The IDMC will then review the next two participants' data before opening the next part of the study (Cohort 2).
  Interventions: Genetic: AXV-101
- Cohort 2 (Experimental): Cohort 2 will include up to nine participants. Participants in this cohort will be administered a therapeutic dose of AXV-101 (5 E11 Vg). The IDMC will review the safety data after each dose for the first three participants, and if no safety concerns are raised, the remaining six participants in cohort 2 will be dosed sequentially.
  Interventions: Genetic: AXV-101

INTERVENTIONS:
Genetic: AXV-101 — This is a gene therapy named AXV-101, being injected into the eye in participants with BBS1 bi-allelic mutations and retinal degeneration. The treated eye will be compared with the eye not injected with AXV-101.

SUMMARY:
The goal of this first in human study is to evaluate the preliminary safety and tolerability of AXV-101 in participants with BBS1. The main questions it aims to answer are:

* Is AXV-101 safe and tolerable to use in participants with BBS1?
* To determine the therapeutic dose of AXV-101 in participants with BBS1
* To investigate the concentration of AXV-101 in blood, urine and tears (both eyes)

Participants will undergo comprehensive ophthalmic assessments to evaluate functional and structural changes from baseline to one year in the treated eye compared with the untreated eye. Additional evaluations will include blood, urine, and tear testing for safety and pharmacokinetics, and quality of life questionnaires completed by both participants and caregivers. Safety will also be assessed by monitoring the frequency and severity of adverse events, including serious adverse events, through medical history, physical examinations, and laboratory testing.

ELIGIBILITY:
To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Male or female participants aged 4 to 17 years (inclusive).
2. Able to provide written informed consent:

   2.1. Parent(s)/guardian(s) prior to the initiation of any study-specific procedures for participants who are under the age of 18 2.2. Participants aged 6-17 years of age may (according to the judgement of the investigator) provide their written assent; consent will also be required from the legal guardian of the participant.

   2.3. Participants aged below 6 years of age will not be required to sign an assent form; however, their views should be considered; consent will be required from the legal guardian of the participant.
3. Participant with a confirmed diagnosis of bi-allelic BBS1 mutations. Molecular diagnosis/genetic testing will have been undertaken by an accredited laboratory using an assay that has the relevant mark of conformity and is used as per its intended use. UK diagnostic genetic laboratories must conform to the Association for Clinical Genomic Science (ACGS) and adopt the ACMG guidelines for the determination of pathogenicity. US diagnostic genetic laboratories must be CLIA-approved.
4. Participants with presentation of retinal degeneration (evidence of early Rod-Cone Dystrophy, Cone-Rod Dystrophy or Night vision loss [nyctalopia])
5. Participants with sufficient viable retinal cells as determined by OCT. Participants must have either:

   5.1. A measurable area of intact ellipsoid within the posterior pole - minimum 1500 microns horizontal width 5.2. ≥3-disc areas of retina without atrophy or pigmentary degeneration within the posterior pole; or 5.3. Remaining visual field within 30 degrees of fixation as measured by a III4e isopter or equivalent.
6. Post-pubertal male participants and female participants of childbearing potential must be willing to comply with the contraceptive requirements

An individual who meets any of the following criteria will be excluded from participation in this trial:

1. A fully blind participant.
2. Participant or participant's legal guardian is unable or unwilling to meet the requirements of the study, or unable to provide written informed consent/assent
3. Participant has been administered any investigational medicinal product (IMP) during the last 6 months prior to individual enrolment of the participant and/or within five half-lives of the previous IMP, whichever is longer
4. Other than as required per protocol, the participant has received immune-modulating agents within 90 days before dosing (use of inhaled corticosteroids to manage chronic respiratory conditions is allowed)
5. Glucocorticoid intolerance
6. Use of other concomitant medications to manage chronic conditions must have been stable for at least 30 days before dosing
7. Presence of severe diabetes or uncontrolled blood glucose
8. Presence of active infection or recent severe infection (elevated WBC)
9. Participant with any prior intraocular surgery in either eye within 6 months
10. Participant with any known sensitivity to AXV-101, its excipients and the medications planned for use in the peri-operative period
11. Participant with significant renal, liver or haematological disease as defined by:
12. Laboratory evidence of liver disease (aspartate aminotransferase greater than two times the upper limit of normal [ULN] of the testing laboratory).
13. Laboratory evidence of renal disease (eGFR<30).
14. Laboratory evidence of haematological disease (absolute neutrophil count < 1,500/mm3; haemoglobin < 0.9 times the lower limit of normal [LLN] of the testing laboratory, by sex; or platelet count < 140,000/mm3).
15. Any pre-existing eye conditions or complicating systemic diseases that would preclude the planned surgery or interfere with the interpretation of the study or the safety of the participant. Active uveitis or intraocular inflammation (infectious or non-infectious). Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function. Examples are malignancies whose treatment could affect central nervous system function (for example: radiation treatment of the orbit; leukaemia with central nervous system (CNS)/optic nerve involvement). Participants with diabetes or sickle cell disease will be excluded if they have had any manifestation of advanced retinopathy (e.g., macular oedema or proliferative changes). Also excluded would be participants with immunodeficiency (acquired or congenital), as there could be susceptibility to opportunistic infection (such as cytomegalovirus retinitis).
16. Participants with evidence of chronic or active viral disease, including:
17. Participant has human immunodeficiency virus HIV-1 or HIV-2, including serological or viral load evidence of HIV 1 or HIV-2.
18. Participant has an active viral infection (systemic bacterial or fungal infection) based on clinical observation.

    18.1. Active hepatitis B (HBV) or C (HCV), and HBsAg, HBcAb, HBV-DNA positivity or HCV-Ribonucleic acid (RNA) viral load positivity, respectively. A negative viral load assay in two samples, collected at least 6 months apart, will be required to be considered negative. Both natural clearers and those who have cleared HCV on antiviral therapy are eligible.
19. Any other circumstance that would not allow the potential participant to complete follow-up examinations during the course of the study or, in the opinion of the Investigator, makes the potential participant unsuitable for the study.
20. Pregnant and/or breastfeeding participant.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the preliminary safety and tolerability of AXV-101 in participants with BBS1 | Through study completion, 5 years
  Evaluation will be via frequency and severity of all adverse events (AEs) including serious adverse events (SAEs) and their relationship to AXV-101 throughout the study (5 years)

SECONDARY OUTCOMES:
To determine the therapeutic dose of AXV-101 in young participants with BBS1 | Change from baseline through 1 year
To investigate the concentration of AXV-101 in blood, urine and tears (both eyes) | From screening to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mariya Moosajee, Principal Investigator — Moorfield Eye Hospital
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided